CLINICAL TRIAL: NCT03280576
Title: Sensitivity and Specificity of Progranulin as a Biomarker for Sepsis
Brief Title: Validation of Progranulin as a Biomarker for Sepsis
Acronym: PROGRANULIN
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: City of Munich (Other Government)
Responsible Party: Principal Investigator, Gustav Schelling,MD, Senior Researcher, Ludwig-Maximilians - University of Munich
Other Study IDs: Progranulin_1
Record Dates: First submitted 2015-11-19; First posted 2017-09-12 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Sepsis
Keywords: Postoperative; Dysfunction Following Cardiac Surgery
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, EDTA blood, blood cells (PAXGENE)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sepsis: Patients with sepsis
- Cardiac Surgery: Patients undergoing cardiac surgery
- Healthy controls: Normal individuals

SUMMARY:
Progranulin blood concentrations in patients with sepsis will be analysed in relation to disease status in order to validate progranulin as a biomarker for sepsis. Patients undergoing cardiac surgery will serve as controls.

DETAILED DESCRIPTION:
Single nucleotide polymorphisms with known effects on Progranulin plasma concentrations will be assessed in a separate analysis. Expression levels of microRNAs isolated from plasma, circulating exosomes and blood cells will be determined by next-generation sequencing to characterize epigenetic influences on progranulin plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis or Septic Shock defined according to SEPSIS-3 criteria - Age > 18 years

Exclusion Criteria:

* No informed consent
* Age < 18 years
* Pregnancy
* Immunosuppression (including transplantation)
* Charlson Comorbidity Index > 0 (healthy volunteers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Sepsis, Patients undergoing cardiac surgery, Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in progranulin plasma concentrations during ICU - therapy | ICU admission, day 1, day 4 of ICU therapy
  Blood samples will be taken at the abovementioned time points

SECONDARY OUTCOMES:
Change in miRNA expression levels in exosomes, serum and blood cells during ICU - therapy | ICU admission, day 1, day 4 of ICU therapy
  Blood samples will be taken at the abovementioned time points

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Schelling, M.D., Principal Investigator — Department of Anaesthesiology LMU
Locations (2):
- Germany (2):
  - Department of Anesthesiology, LMU Munich, Munich, Bavaria
  - Department of Anesthesiology, Klinikum Neuperlach, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brandes F, Borrmann M, Buschmann D, Meidert AS, Reithmair M, Langkamp M, Pridzun L, Kirchner B, Billaud JN, Amin NM, Pearson JC, Klein M, Hauer D, Gevargez Zoubalan C, Lindemann A, Chouker A, Felbinger TW, Steinlein OK, Pfaffl MW, Kaufmann I, Schelling G. Progranulin signaling in sepsis, community-acquired bacterial pneumonia and COVID-19: a comparative, observational study. Intensive Care Med Exp. 2021 Sep 3;9(1):43. doi: 10.1186/s40635-021-00406-7. PMID 34476621